CLINICAL TRIAL: NCT05944263
Title: Effectiveness of an Intervention on Cultivating Character Values of Gratitude, Kindness and Hope to Enhance Mental Well-Being Among Young People in School and Community Settings in India and Nairobi: a Cluster Randomized Controlled Trial
Brief Title: WeRISE: Youth-led Mental Health Transformation Through Cultivating Gratitude, Kindness, and Hope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: citiesRISE (Other)
Collaborators: Schizophrenia Research Foundation (SCARF India) (Unknown); African Population and Health Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TWCF0631
Record Dates: First submitted 2023-06-19; First posted 2023-07-13 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Youth Mental Health
Keywords: adolescents; character strengths; cluster Randomized Controlled Trial (cRCT); co-design; arts based mental health intervention; positive psychology
MeSH Terms: interventions — Acclimatization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The gratitude, kindness and hope (GKH) program (Experimental): This gratitude, kindness and hope (GKH) program will be a structured manual-based intervention that has been adapted and contextualized from the previous work that has been done in this field. Each intervention session will be conducted in the school and community settings by 2 youth trainers aged 18 - 24 and who will be trained in the delivery of the intervention.
  The sessions will be held twice a week, concurrently in schools and in the community. Fifty per cent of the sessions will be supervised by master trainers (who are experts in charge of training the youth trainers on the intervention). The rest of the sessions will be audio-recorded and reviewed randomly during supervision meetings.
  The total duration of each session will be 45 minutes distributed as shown below:
  iv. 5 minutes warm up activity v. 30 minutes practice and explanation of concepts through interactive activities and discussions vi. 10 mins answering questions and designing homework
  Interventions: Behavioral: weRISE; The gratitude, kindness and hope (GKH) program
- The [adapted] Stan Kutcher Teen Mental Health (TMH) program (Active Comparator): The program delivered to the control group is adapted from the Stan Kutcher Teen Mental Health Curriculum. It was initially developed to help enhance the mental health literacy of students and was developed for ages 13 to 15 years which was further adapted for a slightly lower age group (12-14 yrs) as that targeted in this study through simplification of terminologies to ensure age-appropriate content.
  Just like the GKH program, the TMH sessions will be delivered by 2 trained youth trainers in the school and community settings. The program will be delivered over 8 sessions, two sessions a week (i.e. over a span of 4 weeks). Half of the sessions will be supervised by master trainers. Like the GKH program, each session will go for 45 minutes each .
  Interventions: Behavioral: The [adapted] Stan Kutcher Teen Mental Health (TMH) program

INTERVENTIONS:
Behavioral: weRISE; The gratitude, kindness and hope (GKH) program — weRISE is an arts based train the trainer intervention that promotes positive mental health through cultivating gratitude, kindness and hope among youth in schools and informal settlements in India and Kenya
  Arms: The gratitude, kindness and hope (GKH) program
Behavioral: The [adapted] Stan Kutcher Teen Mental Health (TMH) program — The 'Teen Mental Health' curriculum developed by Dr. Stan Kutcher, aims to increase mental health literacy among young people ;will be used in the control group (active comparator group). The control intervention consists of eight sessions (45 minutes each) delivered by older groups of young people (ages 18-24) in schools and community settings through a didactic approach.
  Arms: The [adapted] Stan Kutcher Teen Mental Health (TMH) program

SUMMARY:
The weRISE study's primary aim is to develop and test the effects of an arts-based train-the-trainer intervention developed to cultivate gratitude, kindness, and hope among youth in schools and informal settlements in both India and Kenya, on mental health and well-being outcomes. The core theory of change for weRISE is that through cultivating these key strengths, youth will undergo empowering mindset shifts that equip them to navigate past, present, and future life challenges, including mental ill-health.

Through a cross-country, phased, cluster randomized controlled design, this study will explore the question: what impacts the weRISE intervention has on gratitude, kindness, hope compared with a standard mental health literacy intervention. The investigators will also assess the impacts of weRISE on secondary outcomes such as self-efficacy, the feasibility of the youth-led delivery model, and whether impacts differ depending on setting (schools versus informal settlements, India versus Kenya). The investigators hypothesize that the weRISE intervention will result in greater improvements in mental health and well-being outcomes for youth recipients compared with a standard mental health literacy intervention, and that there will be strong positive relationships between gratitude, kindness, hope, and the mental health and well-being outcomes. The investigators hypothesize that the effects of weRISE will be similar across settings (schools and informal settlements in India and Kenya) and that the youth-led train-the-trainer model will prove effective.

Through this project, investigators will work together with leading experts and youth to develop an overall intervention model, contextualize it for India and Kenya respectively, and package a set of implementation tools for weRISE. Importantly, investigators plan to iterate on the content developed and contextualized for India and Kenya and publish a youth-targeted weRISE guide that will provide any young person anywhere with content and concrete activities. The investigators will also develop a series of academic outputs including scientific articles and conference presentations to disseminate evidence and lessons learned. Finally, the investigators will produce and disseminate a policy brief to facilitate uptake and scaling of weRISE by government officials and other decision-makers.

DETAILED DESCRIPTION:
The adolescent years for young people is a period of crucial life transitions and is fraught with a range of internal and external challenges. Young people in low- and middle-income countries (LMICs) are particularly vulnerable to mental ill health given the exposure to multiple adverse life experiences. Positive psychological interventions have been brought into the social-emotional learning curriculum of western countries and has shown efficacy in supporting the salutary effects of the same in the health and wellbeing of the young people. In most LMICs, where there is less access to psychologists and psychiatrists, the models that are used have only a limited amount of application to the young people who are struggling.

The primary goal of this project is to design and test the effects on mental health and well-being outcomes of an arts-based train-the-trainer intervention, cultivating gratitude, kindness, and hope among youth in schools and informal settlements. The central change theory is that by cultivating these key strengths, youth will experience empowering mind-set shifts that will prepare them to navigate past, present, and future life challenges, including mental illness.

In order to create a robustly tested, adaptable, and scalable intervention that speaks directly to the realities of young people in schools and informal settlements in LMICs, this project will integrate the research currently available in the fields of character development, positive psychology, and mental health. This project will support cross-border collaboration in a number of ways to successfully bridge these rich and diverse sectors. It will bring together specialists from LMICs and high-income countries (HICs), mental health and character development professionals, as well as youth and adult researchers, to produce the fundamental evidence at the nexus of character development and health outcomes.

This project will use a single-blind cluster randomized controlled trial design with 10 clusters 60 young people within schools and 30 in communities recruited from informal settlements in Nairobi and India. The evaluation will employ a mixed methods approach to determine the impact of the intervention on mental wellbeing of young people. Quantitative data will be collected through a survey at baseline and end-line while focus group discussions (FGD) will only be conducted at end-line. These will be analyzed using STATA and NVivo softwares respectively.

This project proposes that, the model and evidence generated will be innovative in a number of ways: 1) it is designed to scale in low-resource settings and takes replicability into account from the start. 2) the intervention's accessibility to a diverse range of youth in LMICs, including the most marginalized, is considered from the start; 3) it departs from the traditional approach of testing interventions based on individual character strengths in order to weave gratitude, kindness, and hope together through an integrated life course (past, present, and future) approach and; 4) the focus is on young people's leadership and their ability to support themselves and their peers. Character strengthening is associated with independent critical thinking inherently required in developing leaders. While this is not an outcome of the study the ability to lead oneself and others with compassion signifies likelihood of a longer-term impact of the character strengthening intervention. Findings from the study would contribute towards improving mental health policies and programs.

ELIGIBILITY:
Inclusion criteria for adolescents in community clusters

* Adolescents between the ages of 12-14 will be recruited in the community matching the demographic of the and living within 5 kilometers of the community-based organization will be recruited
* Parents in the community consent and the adolescent's assent to participate in the program at the community-based organization

Inclusion criteria for adolescents in school clusters

* Students in grade 7-9 in schools that are demographically similar to the community clusters.
* Participating schools and parents in schools provide consent and the adolescents assent to participate in the program at the schools

Inclusion criteria for youth trainers

* Youth trainers should be between the ages 18-24
* Youth trainers' who consent to participate in the program

Exclusion Criteria:

* Young people with forms of disabilities (e.g. sight, intellectual) that make it hard for them to meaningfully participate in the programs will be excluded.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Yes.Participant eligibility is based on self-representation of gender identity.
Enrollment: 840 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Mental health wellbeing | Baseline status of the mental health well-being will be assessed before the intervention. Any change in status of mental health well-being when compared with the baseline will be assessed within 2 weeks and at 2 months post intervention.
  Mental health well-being will be measured using Warwick-Edinburgh Mental Wellbeing Scale. The scale measures aspects of positive affect, functioning and interpersonal relationships as components of wellbeing. The scale has 14 items and scores can range from a minimum of 14 to a maximum of 70 points. Higher scores are associated with higher levels of mental well--being.
Character strengths of gratitude, kindness and hope | Baseline status of the character strengths will be assessed before the intervention. Any change in the character strengths when compared with the baseline will be assessed within 2 weeks and at 2 months post intervention.
  Character strengths of gratitude, kindness and hope have been found to be associated with mental wellbeing and will be measured using the Values in Action Questionnaire (VIA) - Youth Version (25-item questionnaire) among adolescents and youth facilitators.

SECONDARY OUTCOMES:
Depression | Baseline status of depression will be assessed before the intervention. Any change in depression when compared with the baseline will be assessed within 2 weeks and at 2 months post intervention.
  Patient Health Questionnaire - 9 (PHQ - 9) scale will be used to measure depression among adolescents and youth facilitators. It is a short, self-reported, screening tool for the screening of depression in primary care using the Diagnostic and Statistical Manual (DSM)-IV criteria. The PHQ-9 total score ranges from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression)
Anxiety | Baseline status of anxiety will be assessed before the intervention. Any change in anxiety when compared with the baseline will be assessed within 2 weeks and at 2 months post intervention.
  Generalized Anxiety Disorder - 7 (GAD - 7) scale will be used to measure anxiety among adolescents and youth facilitators. It is a 7 item self-reported questionnaire used as a screening tool for measuring generalized anxiety disorder. The GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Moiteryee Sinha, PhD, Principal Investigator — citiesRISE
Locations (2):
- Schizophrenia Research Foundation (SCARF India), Chennai, Tamil Nadu, India
- African Population and Health Research Center (APHRC, Nairobi), Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
This will be updated in due course of time
Supporting Information: Study Protocol, SAP